CLINICAL TRIAL: NCT00166049
Title: A Family Partnership Intervention in Heart Failure
Brief Title: Education and Supportive Partners Improving Self-Care (ENSPIRE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sandra B. Dunbar, RN, Professor, Emory University, Nell Hodgson Woodruff School of Nursing, Emory University
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: IRB00045870; R01NR008800 (NIH); 1R01NR008800-01A1 (NIH)
Record Dates: First submitted 2005-08-31; First posted 2005-09-14 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2013-09

CONDITIONS: Heart Failure
Keywords: Heart failure; Family partnership; Patient family education
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care Attention Control (Placebo Comparator): Usual care with provision of supplemental printed educational material on HF self care
  Interventions: Behavioral: Usual care with educational material
- Group 2 Patient Family Education PFE (Experimental): Patient Family Education PFE Heart Failure Patients and family member dyads were provided with an educational and counseling session, and attended a 2 hour patient-family education session on heart failure self management with emphasis on dietary sodium and medication taking behaviors.
  Interventions: Behavioral: Patient and Family Education; Behavioral: Usual care with educational material
- Group 3 Family Partnership Intervention (Experimental): Patient and family member received one individual dyadic education/counseling session, and two group sessions focused on developing family approaches to HF self management. the emphasis of the two group sessions was on developing autonomy supportive approaches to family support.
  Interventions: Behavioral: Family Partnership Intervention (FPI); Behavioral: Patient and Family Education; Behavioral: Usual care with educational material

INTERVENTIONS:
Behavioral: Family Partnership Intervention (FPI) — HF patient and family receive structured patient and family education sessions plus intervention to improve family communication one month after enrollment.Patient and family member received one individual dyadic education/counseling session after baseline data collection, and two group sessions (2-3 months after baseline) focused on developing family approaches to HF self management.Telephone counseling for the dyad and reinforcing mailed newsletters at 5-6 months after baseline.
  Arms: Group 3 Family Partnership Intervention
Behavioral: Patient and Family Education — HF Patient and one family member receive structured education sessions one month after enrollment.Two sessions, one indivdual with patient-family member dyad after baseline, and one in a group setting between 2-3 months after baseline. The group session was 2 hours in duration. Telephone counseling for the dyad ast 5-6 months, mailed newsletters at Mailed newsletters at 5-6 months.
  Other Names: Patient Family Education PFE
  Arms: Group 2 Patient Family Education PFE; Group 3 Family Partnership Intervention
Behavioral: Usual care with educational material — Usual care with provision of printed educational material, provided once at baseline
  Other Names: Usual Care Attention Control

SUMMARY:
The purpose of the Education and Supportive Partners Improving Self-Care (ENSPIRE) study is to compare the effect of a Family Partnership Intervention (FPI) over patient and family education and usual heart failure care on physical and mental health outcomes over an 8-month period. The study will examine three ways of giving heart failure patients and their family members information. This study will help scientists determine if learning these communication skills will help people with heart failure to better manage their symptoms and improve their health outcomes.

DETAILED DESCRIPTION:
Heart failure is a condition where the heart's pumping ability is reduced, causing shortness of breath, fatigue, fluid-weight gain, and swelling in the abdomen or legs among other symptoms. HF patients can learn to manage their diet, exercise, and medications to reduce these symptoms. Research has shown that people who learn communication skills that involve problem solving and support are often more successful at maintaining lifestyle changes, such as diet and exercise, than those who do not receive this type of training. Routine heart failure care varies, but usually includes patient education about medications and a low sodium diet to prevent fluid buildup and dietary fluid restriction. This study will help advance the scientific understanding of how to best influence and sustain recommended lifestyle changes for HF patients.

The study will investigate three ways of giving HF patients and their family members information. The first method is routine HF care; this serves as the control group. The second method adds a patient and family HF education protocol to routine HF care, and the third method adds a Family Partnership Intervention (FPI). The FPI is an experimental procedure that involves discussion and training in ways to improve communication within families. The study takes place over the course of a year. Two hundred sixty two people and their family members will be asked to participate from Emory, Crawford Long, the VA Medical Center and Grady Healthcare System.

Procedures:

All groups will participate in the following activities:

* Complete questionnaires at start of study, then 4 and 8 months afterward (3 times)
* Keep four appointments lasting 1- 4 hours at the General Clinical Research Center (GCRC) located at Emory or Grady Hospital
* Collect 24-hour urine specimens, one at the start of the study, then 4 and 8 months afterward (3 times)
* Keep a 3-day food record, writing down everything you eat and drink, starting two days before each 24-hour urine collection (3 times)
* Use a medication monitoring system attached to the bottle cap of your heart failure medications
* Take a six-minute walk test in which you walk for up to six minutes at the start of study and then 4 and 8 months afterward (3 times)
* Provide blood samples for Brain Natriuretic Peptide (BNP) levels to determine the level of heart failure present at the start of the study and then 4 and 8 months afterward (3 times)

In addition to the above activities, you will be assigned to one of three groups by a computer program. There is a one in three chance of being in any given group.

First Method: The first group will receive routine HF care in addition to participating in the activities listed above.

Second Method: The second group will attend two HF education classes with their family member and with a registered nurse and dietician in addition to routine HF care and participating in the activities listed above. An educational HF newsletter will be sent and subjects will receive two telephone calls by an RN at two weeks and five months after start of the study (1 time for newsletter and two phone calls).

Third Method: The third group will attend patient and family HF education classes and support group meetings with their family member in addition to routine HF care and participating in the activities listed above. An educational HF newsletter with additional information about building Family Partnerships will be sent and an RN will call at two weeks and five months after start of the study (1 time for newsletter and two phone calls).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of heart failure (New York Heart Association [NYHA] Class II or III)
* Aged 21-79
* Currently taking angiotensin-converting enzyme (ACE) inhibitor and diuretic medications
* Recommended to exercise and low sodium diet
* Willing to participate in educational sessions with a family member
* Willing to spend a minimum of 9 hours and a maximum of 15 hours over an 8-month period
* Willing to travel to either Emory University Hospital or Grady Memorial Hospital General Clinical Research Center (GCRC) for study activities

Exclusion Criteria:

* NYHA Class I or IV heart failure
* Heart attack within the last 6 months
* Kidney failure
* Significant angina/chest pain
* Inability to read and write English

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2005-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Adherence to dietary sodium and medication taking behavior | 4 and 8 months after baseline enrollment.
Physical status: 6-minute walk and brain natriuretic peptide | 4 and 8 months after baseline enrollment.
Psychological status: depressive symptoms | 4 and 8 months after baseline enrollment.
Health related quality of life | 4 and 8 months after baseline enrollment.

SECONDARY OUTCOMES:
Health resource utilization (HRUQ) | 4 and 8 months after baseline enrollment.
Autonomy support (AS) | 4 and 8 months after baseline enrollment.
Perceived family criticism | 4 and 8 months after baseline enrollment.
Knowledge | 4 and 8 months after baseline enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B. Dunbar, RN, DSN, Principal Investigator — Emory University School of Nursing
Locations (4):
- United States (4):
  - Grady Hospital, Atlanta, Georgia
  - Crawford Long Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Veterans Affairs (VA) Medical Center, Decatur, Georgia